CLINICAL TRIAL: NCT06360055
Title: A Prospective, Single-Center, Open-Label Study of the Effect of Oral D-mannose Tablets on the Pharmacokinetics of Dabigatran Etexilate in Healthy Adults
Brief Title: Effect of Oral D-mannose Tablets on Pharmacokinetics of Dabigatranate in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Li Lei, Chief physician, Peking University Third Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: M2024130
Record Dates: First submitted 2024-03-15; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Health
Keywords: D-mannose; Dabigatran Etexilate; P-glycoprotein; pharmacokinetics
MeSH Terms: interventions — Dabigatran; Mannose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-mannose and dabigatran etexilate (Experimental): Subjects will receive a single oral dose of 110mg (low dose specification in the instructions) or lower of dabigatran etexilate on day 1 and day 16 of the trial period. And they will take 3g (1g*3 tablets) of D-mannose tablets every morning and evening from the 2nd day to the 15th day of the trial period, with a total of 6g/day (medium dose specification in the instructions).
  Interventions: Drug: Dabigatran Etexilate; Dietary Supplement: D-mannose

INTERVENTIONS:
Drug: Dabigatran Etexilate — Subjects will receive a single oral dose of 110mg (low dose specification in the instructions) or lower of dabigatran etexilate on an empty stomach on the morning of day 1 and day 16 of the trial period.
  Other Names: Pradaxa
Dietary Supplement: D-mannose — Subjects will take 3g (1g*3 tablets) of D-mannose tablets every morning and evening from the 2nd day to the 15th day of the trial period, with a total of 6g/day (medium dose specification in the instructions).

SUMMARY:
The aim of this study is to investigate the effects of oral D-mannose tablets for 2 consecutive weeks on the pharmacokinetics of dabigatrun etexilate, a P-glycoprotein probe substrate drug, in healthy adults

DETAILED DESCRIPTION:
This study is a prospective, sinale-center, open-label clinical studly, with adult healthy subiects as the research subjects. Healthy adult subjects will receive a single oral dose of 110mg (low dose specification in the instructions) or lower of dabigatran etexilate on day 1 and day 16 of the trial period. Blood samples for dabigatran plasma concentration determination at 0 h(before dosing)2 h, 4 h, 6 h, 12 h and 24 h after dosing will be taken. Subjects will take 3g (1g*3 tablets) of D-mannose tablets every morning and evening from the 2nd day to the 15th day of the trial period, with a total of 6g/day (medium dose specification in the instructions). Blood samples for detection of glycotomic serum concentrations such as D-mannose will be taken 0h before oral administration of dabigatran etexilate on day 1 and 1.5h after oral administration of D-mannose each morning on days 2, 8, and 15 of the trial period.

ELIGIBILITY:
Inclusion Criteria:

1. With full capacity for civil conduct, the age of healthy male subjects is ≥18 years old and ≤45 years old
2. Male weight ≥50 kg; body mass index (BMI) within the range of 19.0~27.0 (including upper and lower limits)
3. Creatinine clearance rate (CRCL: calculated by Cock croft-Gault equation, adult healthy subjects should have CRCL≥90mL/min

Exclusion Criteria:

1. History of fainting of needles and blood.
2. Diseases affecting intestinal P-glycoprotein: severe diarrhea (excretion more than 3 times a day with watery stool characteristics), Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulitis, difficult Identify Clostridium infection (recurrent) or Helicobacter pylori infection.
3. Diabetes mellitus; Impaired fasting glucose (IFG); Impaired glucose tolerance (IGT); Oral hypoglycemic agents (including the use of hypoglycemic agents for weight loss purposes).
4. Diseases or conditions with significant risk of major bleeding, such as current or recent peptic ulcer, malignant neoplasms with high bleeding risk, recent brain or spinal cord injury, recent brain, spinal cord, or eye surgery, recent intracranial hemorrhage, known or suspected Esophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracranial vascular abnormalities.
5. Clinically significant active bleeding.
6. Taking anticoagulants such as unfractionated heparin (UFH), low molecular weight heparin (LMWH) and heparin derivatives (fondaparinux sodium), vitamin K antagonists, rivaroxaban or other direct thrombin inhibitors (recombinant hirudin, bivalirudin); thrombolytic drugs, or current use of antiplatelet aggregation drugs such as GPⅡb/Ⅲa receptor antagonists, ticlopidine, prasugrel, dextran, sulfinpyrazone, aspirin, etc.
7. Use of drugs that may affect the activity of intestinal p-glycoprotein within 1 week before the trial: (1) potent p-glycoprotein inhibitors: amiodarone, verapamil, diltiazem, quinidine, dronedarone, tacrolimus, cyclosporine, protease inhibitors(indinavir, nelfinavir, saquinavir, lopinavir), macrolide antibiotics (erythromycin, clarithromycin, telithromycin, chloramphenicol), azole antifungal drugs (ketoconazole, itraconazole, Posaconazole, voriconazole, fluconazole, miconazole), nefazodone, cobicistat, cimetidine, ciprofloxacin, cyclosporin, fluvoxamine, imatinib, St. John's Wort, ranolazine; (2) Potent P-glycoprotein inducers: rifampicin, carbamazepine, phenytoin, phenobarbital, antiandrogens(enzalutamide, apalutamide), phenobarbital, dexamethasone.
8. Those who have a history of smoking and drinking in the past and who do not agree with the prohibition of smoking and drinking during the trial period: smokers (the average daily cigarettes smoked more than 5 cigarettes within one month before the test); alcoholism: (the average daily drinking within one month before the test≥100mL high-quality liquor/200mL wine / 600mL beer).
9. History of gastrointestinal surgery such as gallbladder or appendectomy, bariatric surgery, etc. within the past 5 years.
10. Positive virological test (human immunodeficiency virus antibody (HIV-Ab), syphilis serological test, hepatitis B virus surface antigen (HBsAg) or hepatitis C virus antibody (HCV-Ab)) within 6 months before screening.
11. Those who have participated in clinical trials of any dug or medial device within 6 months before screening (in the case of drug clinical trials those who participated in the previous clinical trial before screening have more than 5 half-lives).
12. Subjects who are considered by the investigator to have any factors that are not suitable for participating in this trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of dabigatran | 0 hours before and 2, 6, 10 and 24 hours after administration of dabigatran etexilate on the day 1 and day 16 of the trial period.
  Plasma concentration of dabigatran will be measured by liquid chromatography-tandem mass spectrometry
Serum concentrations of glycoomics such as D-mannose | 0 hours before administration of dabigatran etexilate of day 1 and 1.5 hours after D-mannose administration in the morning of day 2, day 8 and day 15.
  Serum concentrations of glycoomics such as D-mannose will be measured by gas chromatography-tandem mass spectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marzolini C, Paus E, Buclin T, Kim RB. Polymorphisms in human MDR1 (P-glycoprotein): recent advances and clinical relevance. Clin Pharmacol Ther. 2004 Jan;75(1):13-33. doi: 10.1016/j.clpt.2003.09.012. PMID 14749689
- [Background] Elmeliegy M, Vourvahis M, Guo C, Wang DD. Effect of P-glycoprotein (P-gp) Inducers on Exposure of P-gp Substrates: Review of Clinical Drug-Drug Interaction Studies. Clin Pharmacokinet. 2020 Jun;59(6):699-714. doi: 10.1007/s40262-020-00867-1. PMID 32052379
- [Background] Dong L, Xie J, Wang Y, Jiang H, Chen K, Li D, Wang J, Liu Y, He J, Zhou J, Zhang L, Lu X, Zou X, Wang XY, Wang Q, Chen Z, Zuo D. Mannose ameliorates experimental colitis by protecting intestinal barrier integrity. Nat Commun. 2022 Aug 16;13(1):4804. doi: 10.1038/s41467-022-32505-8. PMID 35974017